CLINICAL TRIAL: NCT03489551
Title: Feasibility of Prophylactic Haldol to Prevent Delirium in Cancer Patients
Acronym: PHDC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michelle Weckmann (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Michelle Weckmann, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201107736
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Stem Cell Transplant Complications; Delirium
MeSH Terms: conditions — Delirium | interventions — Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Haldol in patients undergoing HSCT (Experimental): Prior to stem cell transplant participants will receive 5mg of liquid or pill form, oral Haldol. Every other day visits will take place following the first administration of the study drug until 14 days after the transplant.
  Interventions: Drug: Haldol

INTERVENTIONS:
Drug: Haldol
  Other Names: haloperidol

SUMMARY:
This research study proposes to conduct an open label, feasibility study administering prophylactic oral haldol to patients undergoing a hematopoietic stem cell transplant (HSCT).

The study will address the following research aims: 1) To demonstrate the feasibility of enrolling HSCT patients in a prophylactic medication trial, 2) To determine the tolerability of oral haldol in HSCT patients and 2) To compare rates of delirium in HSCT patients who receive prophylactic haldol with an untreated historical control group.

DETAILED DESCRIPTION:
This is an open label, safety & feasibility, clinical drug trial. We will use historical controls from previous research with bone marrow transplant patients and delirium incidence at University of Iowa Hospitals and Clinics (UIHC) to evaluate the efficacy of prophylactic Haldol in the prevention of delirium. This study will recruit adult cancer patients undergoing hematopoietic stem cell transplant (HSCT) at UIHC.

ELIGIBILITY:
Inclusion Criteria:

* The participant must undergo an autologous or allogeneic bone marrow or stem cell transplant
* The participant is 18 years of age or older
* The participant provides written consent

Exclusion Criteria:

* The participant has a QTc of >450 msec at the time of enrollment
* The participant used any antipsychotic medications within the last 30 days
* The participant has any significant allergies or past intolerance to Haloperidol
* The participant has a history of major neurological, metabolic, psychiatric, or cardiovascular disease, cerebrovascular event, or substance abuse
* The participant has a history of mental retardation or learning disability that, at the discretion of the investigator, could affect their ability to complete study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Weckmann, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Haldol in Patients Undergoing HSCT: Prior to stem cell transplant participants will receive 5mg of liquid or pill form, oral Haldol. Every other day visits will take place following the first administration of the study drug until 14 days after the transplant.
  Haldol
Period: Overall Study
Arm/Group | Oral Haldol in Patients Undergoing HSCT
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 15 participants completed treatment
Arm/Group | Oral Haldol in Patients Undergoing HSCT
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [46.8 to 70.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Side Effects and Tolerability of Haldol in Patients With Undergoing Hematopoietic Stem Cell Transplant
Description: Categorize and quantify adverse events from start of drug (day 1) to end of study drug per (CTCAE) version 4.0
Time Frame: Daily, up to 14 days following transplant
Population: Participants completing treatment
Measure: Number; unit: Adverse Event
Arm/Group | Oral Haldol in Patients Undergoing HSCT
Number analyzed (Participants) | 15
Adverse Event | 1

ADVERSE EVENTS:
Arm/Group | Oral Haldol in Patients Undergoing HSCT
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Haldol in Patients Undergoing HSCT (N=15)
Excessive sedation (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes